CLINICAL TRIAL: NCT05463991
Title: Bioengineered Collagen Scaffold Implant as an Alternative to Conventional Buccal Mucosa for Substitution Urethroplasty of Distal Urethral Strictures. - A Pilot Stud
Brief Title: Bioengineered Collagen Implant for Urethral Stricture Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regenosca SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FIH-BCI
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bioengineered collagen implant (Experimental): Standard technique of doing a substitution urethroplasty with no modification to the surgical steps. Instead of an autologous oral bucal mucosa graft, the bioengineered collagen implant is sutured to the healty urethral area after incision of the urethra at the stricture location.
  Interventions: Device: Bioengineered collagen implant

INTERVENTIONS:
Device: Bioengineered collagen implant — Urethral stricture repair

SUMMARY:
The field of research for this study is tissue engineering and the utilization of a bioengineered collagen implant as a substitute biomaterial for conventional buccal mucosa in substitution urethroplasty of distal urethral strictures.

DETAILED DESCRIPTION:
Urethral stricture is defined as the abnormal narrowing of the urethral lumen in the area of the corpus spongiosum. A stricture is the result of ischemic spongiofibrosis manifesting as scar tissue in the corpus spongiosum. Long-term consequences are chronic fistulation through the skin, recurrent sepsis, bladder stones, obstructive uropathy, obstructive nephropathy, and finally renal failure.

Current available surgical techniques for urethral stricture repair require harvesting of grafts from autologous sites resulting in additional risks of complications at the tissue harvest site and additional pain to the patient.

The hypothesis of this study is that the developed bioengineered collagen implant can be used as an alternative biomaterial to buccal mucosa for substitution urethroplasty in urethral stricture patients.

ELIGIBILITY:
Inclusion Criteria:

Adult males with urethral stricture less than 3 cm (anywhere from penile to bulbar urethra not including the membranous urethra) with existing lumen of at least 6 Fr suitable for augmentation urethroplasty. The stricture may be due to trauma or infection.

Exclusion Criteria:

* Known bovine collagen allergy
* Current urinary tract infection
* Chronic renal failure
* Diabeted
* Neurological diseases
* Chronic obstructive pulmonary diseases
* Sleep disturbances
* Depression
* Former cancer treatment
* Smokers
* Recurrent stricture

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Urethral patency | four weeks post-surgery
  A peri-urethrogram will be performed prior to catheter removal.

SECONDARY OUTCOMES:
Voiding symptoms | two months up-to twenty-four months post-surgery
  Participants are filling out the International Prostate Symptom Score (IPSS) questionnaire.
Urine flow | two months up-to twenty-four months post-surgery
  Participants are undergoing an uroflowmetry. This test measures the volume of urine released from the body, the speed with which it is released, and how long the release takes.

CONTACTS AND LOCATIONS:
Overall Officials: Teng Aik Ong, Prof, Principal Investigator — University of Malaya Medical Center
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No